CLINICAL TRIAL: NCT05686616
Title: Multicenter, Randomized, Controlled Trial to Assess the Efficacy of Sodium Glucose Cotransporter-2 Inhibitor add-on Treatment in Patients With Severe Tricuspid Regurgitation
Brief Title: SGLT2 Inhibitor for Severe Tricuspid Regurgitation
Acronym: Reduction-TR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Ji Park, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reduction TR
Record Dates: First submitted 2023-01-09; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Tricuspid Regurgitation
Keywords: tricuspid regurgitation; SGLT2 inhibitor
MeSH Terms: conditions — Tricuspid Valve Insufficiency | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2 inhibitor group (Active Comparator): Participants will take dapagliflozin propanediol hydrate 12.3 mg once a day for a total of 48 weeks.
  Interventions: Drug: Dapagliflozin Propanediol Hydrate 12.3 mg
- Conventional treatment group (No Intervention): Participants will continue the existing medications for severe TR.

INTERVENTIONS:
Drug: Dapagliflozin Propanediol Hydrate 12.3 mg — Forxiga 10mg will be added on the conventional treatment for SGL2 inhibitor group.
  Other Names: Forxiga Tablet 10mg
  Arms: SGLT2 inhibitor group

SUMMARY:
The purpose of this study to identify the efficacy of sodium glucose cotransporter 2 inhibitors add-on treatment on right ventricular remodeling and the amount of severe tricuspid regurgitation (TR) in patients with isolated severe TR.

DETAILED DESCRIPTION:
After being informed consent about the study and potential risk, all patients giving written informed consent will undergo a 1 month screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in an open-label manner in a 1:1 ratio to SGLT2i add-on group or conventional treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Participant over 20 years of age who understands the research protocol and has written informed consent
2. Participant with severe tricuspid valve regurgitation

   * Vena contracta width > 0.7cm or effective regurgitant orifice (ERO)≥40mm2 for more than 1 month despite medical treatment
   * Participant with left ventricular ejection fraction ≥ 40%
   * Participant with NYHA class II or more

Exclusion Criteria:

1. Patient with severe mitral valve or aortic valve disease
2. Left ventricular ejection fraction less than 40%*
3. Patient with severe pulmonary hypertension (TR Vmax > 4m/s)
4. Patient with acute heart failure or dyspnea of NYHA functional class IV or higher
5. Symptomatic hypotension or systolic blood pressure < 90 mmHg at screening
6. Patient with severe lung disease (asthma, obstructive pulmonary disease, acute pulmonary embolism)
7. Patients with renal failure (Estimated GFR < 30 mL/min/1.73 m2) or on dialysis
8. Patient with Type 1 diabetes
9. If a woman of childbearing potential has not used double contraception
10. Patients with claustrophobia or with metallic implants unsuitable for magnetic resonance imaging
11. Blood AST or ALT value is more than twice the upper limit of normal or symptoms and signs of cirrhosis (history of hepatic coma, history of esophageal varices, history of symptomatic ascites)
12. Life expectancy is less than one year
13. Patient who already take SGLT-2 inhibitor
14. A history of hypersensitivity or allergy to SGLT2 inhibitor

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-04-13 (Estimated); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Difference of RVESVi by CMR from baseline to 12 months follow-up (∆RVESVi) | Baseline and month 12
  RVESV index at 12 months - RVESV index at baseline

SECONDARY OUTCOMES:
Difference of RVEDVi by CMR from baseline to 12 months follow-up (∆RVEDVi) | Baseline and month 12
  RVEDV index at 12 months - RVEDV index at baseline
Difference of RV ejection fraction by CMR from baseline to 12 months follow-up (∆RVEF) | Baseline and month 12
  RVEF at 12 months - RVEF at baseline
Difference of Vena contracta width of TR by echocardiography from baseline to 12 months follow-up (∆VCW) | Baseline and month 12
  TR VCW at 12 months - TR VCW at baseline
Difference of TV annulus diameter by echocardiography from baseline to 12 months follow-up | Baseline and month 12
  Tricuspid annulus diameter at 12 months - Tricuspid annulus diameter at baseline
Difference of TR volume by CMR from baseline to 12 months follow-up | Baseline and month 12
  TR volume at 12 months - TR volume at baseline

OTHER OUTCOMES:
Occurrence of cardiovascular death or hospitalization for right heart failure* during 12 months | 12 months after enrollment
  development of cardiovascular death or admission for heart failure
Occurrence of tricuspid valve surgery during 12 months | 12 months after enrollment
  TV surgery
Difference of NT-proBNP from baseline to 12 months follow-up | Baseline and month 12
  NT-proBNP at 12 months - NT-proBNP at baseline
Occurrence of renal dysfunction (creatinine > 2mg/dL) | 12 months after enrollment
  Newly developed renal dysfunction during follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Sung Ji Park, MD, PhD, Principal Investigator — Heart Vascular Stroke Institute, Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea